CLINICAL TRIAL: NCT07011641
Title: Parental Burnout - Checking the Effectiveness of Therapeutic Interventions Based on the Basics of Cognitive-behavioral Therapy
Brief Title: Parental Burnout Interventions
Acronym: PBA-INT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Maria Grzegorzewska University, Warsaw (Other)
Responsible Party: Principal Investigator, Dawid Scigala, PhD, The Maria Grzegorzewska University, Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBA2021; CONSENT NO. 27/2021 (Other: The Senate Committee on Research Ethics of the Maria Grzegorzewska University in Warsaw)
Record Dates: First submitted 2025-05-31; First posted 2025-06-09 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Parental Burnout

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- Intervention group (Experimental)
  Interventions: Behavioral: Structured Online CBT Program

INTERVENTIONS:
Behavioral: Structured Online CBT Program — The interventions consisted of eight weekly group sessions (1.5-2 hours each), with each session addressing a specific theme identified through literature as closely related to parental burnout. The sequential themes were the social pressure on parenting, the dynamic balance of parental stressors and resources, parental perfectionism, personal emotional competencies, parent-child relationship quality, co-parenting quality, help seeking, with a last session focused on relapse prevention.
  Arms: Intervention group

SUMMARY:
This interventional, retrospective study evaluated the effectiveness of online therapeutic interventions based on basic principles of cognitive-behavioral therapy (CBT) in reducing parental burnout. A total of 60 participants took part in the study conducted entirely online between June 2021 and September 2022. The primary objective was to determine whether a structured intervention, designed specifically for this project, could significantly reduce the levels of burnout experienced by parents. The interventions were delivered remotely and did not involve any pharmacological treatment. The study was conducted after obtaining ethical approval and is being registered retrospectively to ensure transparency and research accessibility.

DETAILED DESCRIPTION:
Procedure Following initial screening interviews, parents were randomly assigned to one of four groups of 15 participants each. Two groups immediately received the intervention, while the other two groups served as waiting-list controls, did not participate in the intervention in the described study, but constituted the control group. Mothers in control groups were monitored for burnout levels with the use of the Parental Burnout Assessment (PBA) and were offered the opportunity to receive the intervention six months after their enrolment.

The group-based therapeutic intervention (see below for the detail of the intervention) was delivered to two groups of parents online, while the third and fourth groups were control groups.

After completing an online application form, each parent had a brief online meeting with a psychologist to assess the eligibility criteria, i.e.: having at least one child still living at home, experiencing symptoms of parental burnout, and being motivated to participate in therapeutic interactions. During the meeting, parents were asked to explain their reasons for wishing to join the group. On that basis, parents whose expectations did not relate to the reduction of parental burnout symptoms (e.g., improvement of a disabled child functioning) were excluded. Due to the fact that parental burnout increases the risk of suicide, all persons who volunteered for the project were diagnosed in this respect during the first individual meeting with a psychologist, and were invited to the first intervention group, if the risk of suicidal thoughts or tendencies appeared.

After the online consultation, the method for delivering the parental burnout questionnaire and the informed consent form was established. These documents were provided in paper form and subsequently returned by the participants to the study author. The content of the informed consent form was approved by the Ethics Committee, and the entire procedure was conducted in accordance with the 1964 Declaration of Helsinki. The study was conducted in accordance with the recommendations of the Research Ethics Committee of the Maria Grzegorzewska University in Warsaw (Consent No. 27/2021).

All signed an informed consent form and were advised of their right to withdraw from the study at any time. To ensure data confidentiality, participants were identified by means of anonymous codes. The eligible parents were randomly assigned to four groups (1- intervention, 2- intervention, 3-control and 4-control). Only those who exhibited suicidal thoughts / tendencies or scored more than 53 points on the PBA questionnaire, which suggest high degree of parental burnout were given priority to the intervention group. However, in this study none of the parents revealed any suicide risk. In order to comply with all ethical standards, those in the control groups were given an opportunity to participate in a free of charge intervention after the final stage of the study, like the other groups. Parents were assessed three times: T1 baseline, T2 post-intervention or equivalent timing for controls and T3 six-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

Adult (18 years or older)

Has at least one child currently living at home

Reports experiencing symptoms of parental burnout

Willing and motivated to participate in an online therapeutic intervention

Has access to a device with internet connectivity

Exclusion Criteria:

* Current diagnosis of a severe psychiatric disorder (e.g., psychosis, bipolar disorder)

Currently receiving psychological therapy targeting parental burnout

Inability to understand and communicate in the language of the intervention

No access to stable internet or a suitable device

Participation in another clinical trial during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Parental Burnout as measured by the Parental Burnout Assessment (PBA) | From baseline to month 6 (end of intervention)
  Change in total scores on the Parental Burnout Assessment (PBA) from baseline to the end of the 8-week online intervention. Higher scores reflect greater parental burnout. The scale includes emotional exhaustion, contrast with previous parental self, emotional distancing, and feelings of being fed up.

CONTACTS AND LOCATIONS:
Locations (1):
- The Maria Grzegorzewska University in Warsaw, Warsaw, Poland, Poland

IPD SHARING:
Plan to Share IPD: Undecided